CLINICAL TRIAL: NCT02317692
Title: Standard Versus Culturally-Modified ADHD Treatment
Brief Title: ADHD Treatment for Latino Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Alyson Gerdes, Associate Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR-2871
Record Dates: First submitted 2014-12-09; First posted 2014-12-16 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard ADHD parent training (Active Comparator): 8 sessions of evidence-based parent training plus school intervention
  Interventions: Behavioral: Parent training
- Culturally-modified ADHD parent training (Experimental): 8 sessions of culturally-modified parent training plus school intervention
  Interventions: Behavioral: Parent training

INTERVENTIONS:
Behavioral: Parent training

SUMMARY:
The current pilot study aims to close the existing gap in our knowledge about effective psychosocial treatments for Latino families by providing preliminary data regarding the acceptability and efficacy of a culturally-modified ADHD treatment and possible moderators that will support a future R01. Specifically, the current pilot study is the first step in a larger program of research aimed at definitively determining if culturally-modified ADHD treatment outperforms standard treatment when examining engagement and acceptability outcomes, as well as symptomatology and parental functioning, and if so, which treatment modifications are necessary and for whom. The following study aims will be examined.

1. Aim 1 is to explore if the culturally-modified treatment results in better engagement and acceptability outcomes (i.e., parental attendance, retention, engagement, and satisfaction) than standard treatment and to determine the strength of these effects.
2. Aim 2 is to explore if the culturally-modified treatment results in improvements in ADHD symptomatology, as well as parental functioning (i.e., parenting stress and efficacy), to explore if the modified treatment results in similar or greater improvements than standard treatment, and to determine the strength of these effects.
3. Aim 3 is to explore possible moderators (i.e., socioeconomic status (SES) and behavioral and cognitive acculturation) that may explain the relationship between treatment type (i.e., standard versus culturally-modified) and outcomes and to determine the strength of these interactions.

ELIGIBILITY:
Inclusion Criteria:

* Children must

  1. Self-identify as Latino and be between the ages of 5 and 13 years at the time of the initial assessment
  2. Receive a primary diagnosis of ADHD
  3. If medicated for ADHD, be on a stable dose of medication for at least two weeks prior to the assessment
* Participating parents must

  1. Self-identify as Latino
  2. Be fluent in Spanish
  3. Be able and willing to provide informed consent and comply with the study procedures, including being assigned either to standard or culturally-modified treatment
  4. Have no immediate plans to pursue other treatment for their child's ADHD or to change their child's medication (if already medicated) over the next eight weeks

Exclusion Criteria:

* Children must not meet DSM-5 diagnostic criteria for Intellectual Disability, Autism Spectrum Disorder, or a psychotic disorder

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of participants includes children, mothers, and fathers.
Pre-assignment Details: 1 father did not complete post-treatment measures.
Units Other Than Participants: Families
Groups:
- Standard ADHD Parent Training: 8 sessions of evidence-based parent training plus school intervention
  Parent training
- Culturally-modified ADHD Parent Training: 8 sessions of culturally-modified parent training plus school intervention
  Parent training
Period: Overall Study
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Started | 69; 30 Families | 77; 31 Families
Completed | 63; 27 Families | 77; 31 Families
Not Completed | 6; 3 Families | 0; 0 Families

BASELINE CHARACTERISTICS:
Units Other Than Participants: Families
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training | Total
Number analyzed (Participants) | 69 | 77 | 146
Number analyzed (Families) | 30 | 31 | 61
Age, Continuous [Mean (Full Range); unit: years] — Population: Data on age were only collected for children.
  years
    number analyzed (Participants) | 30 | 31 | 61
    (all) | 8.13 [5 to 12] | 7.84 [5 to 13] | 7.98 [5 to 13]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only includes data from children.
  Participants
    number analyzed (Participants) | 30 | 31 | 61
    Female | 9 | 8 | 17
    Male | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data only represents children.
  Participants
    number analyzed (Participants) | 30 | 31 | 61
    Hispanic or Latino | 30 | 31 | 61
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Families]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Treatment - Treatment Completion (Number of Families Who Completed Treatment)
Description: Number of families who completed treatment (recorded by clinician)
Time Frame: 8 weeks
Measure: Count of Units; unit: Families
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 69 | 77
Number analyzed (Families) | 30 | 31
Families | 27 | 31

2. Primary Outcome: Engagement in Treatment - Sessions Attended
Description: Number of sessions attended by each family (recorded by clinician)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 69 | 77
Number analyzed (Families) | 30 | 31
sessions | 6.93 (1.46) | 7.52 (.93)

3. Primary Outcome: Engagement in Treatment - Homework Completion (% of Completed Homework)
Description: (recorded by clinician - homework was assigned every week and was expected to be returned at the next week's session)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of completed homework
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 69 | 77
Number analyzed (Families) | 30 | 31
percentage of completed homework | 68.95 (24.36) | 88.83 (13.63)

4. Primary Outcome: Acceptability of Treatment (Summary Score of Therapy Attitude Inventory)
Description: Parental report of satisfaction with treatment (summary score of Therapy Attitude Inventory) Range=10-50; higher scores represent greater satisfaction (a better outcome)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 63 | 77
Number analyzed (Families) | 27 | 31
units on a scale | 44.74 (3.57) | 46.93 (3.17)

5. Secondary Outcome: Change in ADHD Symptoms (Inattention Subscale of Disruptive Behavior Disorders Rating Scale)
Description: Pre-treatment to post-treatment change on inattention subscale of Disruptive Behavior Disorders Rating Scale (completed by parent) Range=0-3; the larger the number, the greater the symptoms Difference in mean pre and post scores for each group, so SD was not calculated.
Time Frame: Baseline to 8 weeks
Measure: Number; unit: units on a scale
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 63 | 77
Number analyzed (Families) | 27 | 31
units on a scale | -.14 | -.44

6. Secondary Outcome: Change in Parental Functioning (Maternal Parenting Stress)
Description: Pre-treatment to post-treatment change on summary score of Parenting Stress Index-Short Form (completed by mothers) Range=0-144; the larger the number, the greater stress Difference in mean pre and post scores for each group, so SD was not calculated.
Time Frame: 8 weeks
Population: Only mothers completed.
Measure: Number; unit: units on a scale
Units Other Than Participants: Families
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 27 | 30
Number analyzed (Families) | 27 | 30
units on a scale | -7.22 | -11.1

7. Secondary Outcome: Effects of Socioeconomic Status and Parental Acculturation on Treatment Outcomes (Parental Report)
Description: Socioeconomic status computed based on parental report of education and occupation (assessed on demographic form). Acculturation based on parental report on the Acculturation Rating Scale for Mexican Americans-II and the Mexican American Cultural Values for Adolescents and Adults.
Time Frame: 8 weeks
Population: We did not examine this outcome measure due to a lack of variability on the SES and acculturation measure.
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard ADHD Parent Training | Culturally-modified ADHD Parent Training
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/77
Other Adverse Events (participants affected / at risk) | 0/69 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No